CLINICAL TRIAL: NCT00728325
Title: The Impact of Supported Employment Versus Standard Vocational Rehabilitation in Veterans With PTSD
Brief Title: Impact of Supported Employment Versus Standard Vocational Rehabilitation in Veterans With Post-traumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lori Davis, MD, ACOS Research and Development, Tuscaloosa Research & Education Advancement Corporation
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PT074312; VA IRB ID: 00123
Record Dates: First submitted 2008-07-15; First posted 2008-08-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: PTSD
Keywords: PTSD; Vocational Rehabilitation; Supported Employment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Employment, Supported

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard Vocational Rehabilitation (VRP)
  Interventions: Behavioral: Standard Vocational Rehabilitation (VRP)
- 2 (Experimental): Supported Employment (SE)
  Interventions: Behavioral: Supported Employment (SE)

INTERVENTIONS:
Behavioral: Supported Employment (SE) — SE(IPS)involves: a vocational rehabilitation employment specialist who is integrated into the clinical treatment team, carries out all phases of the vocational services, provides predominantly community-based services, provides assertive engagement and outreach, has a case load of ≤ 25 clients; engages in rapid job search, individualized placement in diverse and potentially permanent competitive job(s), ongoing work-based vocational assessment, and assistance in finding subsequent jobs if needed with the view that all jobs are positive learning experiences; continuous time-unlimited follow-along supports to provide vocational services; and weekly group supervision with IPS/VRP team and with IPS supervisor/trainer monthly.
  Other Names: Veterans in Vocational Rehabilitation Program
  Arms: 2
Behavioral: Standard Vocational Rehabilitation (VRP) — Standard Vocational Rehabilitation (VRP) includes 1) the Vocational Assistance Program (includes routine prevocational testing and evaluation for all patients upon referral to VRP), 2) Vocational Rehabilitation Therapy that operates under the Compensated Work Therapy/Veterans Industries (CWT) and provides a work regimen with monetary incentives derived from contracts whereby participants are paid on a piece rate basis related to their production, and 3) Transitional Work Program (TWP) that includes a temporary work experience either within the VAMC or in community settings (called the Transitional Work External or TWE).
  Other Names: Veterans in Vocational Rehabilitation Program
  Arms: 1

SUMMARY:
This prospective randomized study evaluates the impact of Supportive Employment (SE) compared to standard vocational rehabilitation (VRP) on occupational, sobriety, psychiatric, and quality of life outcomes and health care costs for veterans with chronic posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Hypotheses or Key Questions

I. Primary Hypothesis (obtained + maintained employment): Subjects assigned to IPS will have a higher maintained employed rate for the 12-mo observation period than their standard VRP counterparts.

* I.a. First Component Primary Hypothesis (obtained employment): Subjects assigned to IPS will have higher rates of obtained employment for the 12-mo observation period than the VRP subjects.
* I.b. Second Component Primary Hypothesis (maintained employment): Among those subjects employed, those assigned to IPS will have worked more weeks for the 12-mo observation period than the VRP subjects.

II. Secondary Hypothesis: Those subjects who obtain competitive employment will have significantly reduced symptoms of PTSD from baseline to endpoint compared to those subjects who do not obtain competitive employment.

III. Confirmatory and Correlational Hypotheses: Compared to VRP subjects, those subjects assigned to IPS will have:

* greater work intensity (# weeks, days, # hours, wages earned)
* higher total earnings
* greater improvement in quality of life outcomes

Supplemental hypothesis (moderator): Because of the superior integration with the mental health (MH) treatment team, social work services, and community resources that the IPS-SE employment specialist provides as part of this model, we hypothesize that the IPS-SE model will have greater success in the maintenance of competitive employment compared to standard VRP for veterans with PTSD challenged in one or more of these psychosocial domains. From a research perspective, a variable that characterizes subjects for whom a particular treatment will be effective is called a moderator of treatment.

The hypothesized moderators of IPS-SE and standard VRP for subjects with PTSD are: 1) Transportation, 2) Housing, 3) Financial Means, and 4) Family Care Burden. We hypothesize that these variables will have moderating effects for each of two outcomes: 1) number of weeks the participant is competitively employed during the 12-month study period and 2) their score on the Sheehan Disability Scale.

Several principles are important in defining a moderator. First, the moderator must precede treatment. In our RCT, these psychosocial domains are baseline characteristics of subjects enrolled in the study. Second, the moderator must be uncorrelated with treatment choice. This will be the case in this RCT due to a 1:1 randomization, which should balance baseline characteristics between the two groups. Third, a moderator of treatment must have a differential effect of treatment for each level of the moderator. The treatment effect (e.g., active vs. comparator) must be shown to be greater for one level of the moderator (i.e. IPS-SE will show a greater effect size than standard VRP in subjects with a moderator present). Also, an index that combines these domains will be explored and formulated to identify subjects that may benefit to greater extent from IPS-SE.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* diagnosis of PTSD (based on MINI)
* male or female
* any race or ethnicity
* age 19-60
* currently unemployed
* interested in competitive employment
* planning to remain in a 100-mile radius of participating VAMC for the 12- mo duration

Exclusion Criteria:

* Lifetime history of severe traumatic brain injury that has resulted in severe cognitive disorder
* diagnosis of schizophrenia, schizoaffective disorder, or bipolar I disorder
* dementia (a standard exclusion from VRP)
* immediate need of detoxification from alcohol or drugs (a standard VRP exclusion)
* pending active legal charges or expected incarceration

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Using an intent to treat analysis, subjects' maintained employed rate is measured using the Employment Index. | 12 months

SECONDARY OUTCOMES:
Using an intent-to-treat analysis, the change from baseline to endpoint in PTSD symptoms is compared between groups using the Clinician Administered PTSD Scale (CAPS). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori L. Davis, M.D., Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - Bedford VA Medical Center, Bedford, Massachusetts